CLINICAL TRIAL: NCT01866852
Title: The Formation of Healthy, Stable Romantic Relationships During Young Adulthood: A Developmental and Dyadic Perspective
Brief Title: Expansion of Childhood Relationship Study to Young Adult Romantic Relationships
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913113; 13-CH-N113
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-12-19

CONDITIONS: Healthy
Keywords: Longitudinal Study; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

- An earlier study on child development focused on the relationship between children and their caregivers (usually mothers). It looked at how this relationship influenced children's social and mental development. It also studied how these children related with family members and friends. Researchers are now interested in expanding the study with the same group of children. They want to look at these children, who are now young adults, and focus on their current romantic relationships. This new study will look at how child development affects the formation of stable, mature romantic relationships in young adulthood. Original child study participants and their significant others will be included in the new study. Only participants who are living together with a partner will be studied.

Objectives:

- To look at romantic partnerships in a childhood study s original participants and their significant others.

Eligibility:

* Participants of the 88-CH-32 study who are at least 18 years of age.
* Significant others of the study participants who are at least 18 years of age.
* Original participants and significant others must be cohabiting (living together).

Design:

* No screening tests will be required for this study. No study visits will be needed. Samples will not be collected.
* Original study participants will fill out four online questionnaires. They will be on a National Institute of Child Health and Human Development (NICHHD) website. They will ask personal questions about relationships with the current romantic partner and other important people. The questions will take about 25 minutes to answer.
* Significant others will fill out 13 online questionnaires. They will be on a NICHHD website. They will ask personal questions about the romantic partner and other important people. The questions will take about 1.5 hours to answer.
* All participants will receive a small amount of money for completing the study.

DETAILED DESCRIPTION:
The purpose of this study is to expand our ongoing longitudinal study (study 88-CH-32) by gathering information about romantic partnerships from both the longitudinal study s now young adult target children, who were 5 months old when the study began and are now as old as 23 years of age, and their significant others. Because the target children are approaching the age when they form lasting romantic relationships, we wish to track these partnerships as they form. With these data, we will be uniquely suited to identify how key individual and inter-personal factors at distinct points of development (i.e., childhood, adolescence, and young adulthood) influence the formation of stable, emotionally intimate, mutually dependent romantic relationships during young adulthood. In particular, we aim to disentangle the influence of childhood and adolescent interpersonal experiences in other relational spheres (i.e., relationships with parents and friends) from the influence of contemporary characteristics of both members of the romantic dyad. As part of our examination, in addition to relationship quality, we focus on the strength of each dyad member s attachment to his or her parents as well as each other, thereby allowing for the examination of attachment transfer, an important yet understudied characteristic of successful romantic relationship formation.

Only cohabiting (whether married or otherwise) young-adult romantic dyads that include a target child from our existing longitudinal study (dyad N equals 250; 500 young adults overall, all volunteers) will be eligible to participate in this new data collection. By limiting eligibility in this way, we will have data extending back to infancy for one member of each young-adult romantic dyad. All data collected will be collected via a secure, password-protected website.

As part of our on-going longitudinal study, we already collected (or will collect) individual information from the young adult target children (mental health, attachment style, attachment strength, personality, substance use). We propose here to collect complementary individual information from the significant others of young adult target children as well as dyad-level information (relationship satisfaction and household functioning) from both members of the cohabiting romantic dyad. Combined with existing data from our longitudinal study, these new data will enable us to move beyond most current research focused on the developmental antecedents of successful young adult romantic relationships and examine how an individual s past interpersonal experiences interplay with the contemporary characteristics of both young-adult romantic dyad members to influence the state of the romantic dyad.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Among the young adult target children from study 88-CH-32 (N = 250), those with significant others are eligible to participate in this study, as are their significant others. However if a target child s significant other is a minor (i.e., under the age of 18), that significant other will not be eligible to participate.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Original child (now adult) study participants from protocol 88-CH-0032 and their significant others will be included in the new study. Only participants who are living together with a partner will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2013-05-29; Primary Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Romantic Relationship Quality | Ongoing
  Romantic Relationship Quality

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Putnick, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
All data will be stored permanently in an archival database by the National Institutes of Health. No one other than members of the research team will have access to the data without the explicit consent of the volunteer adult.

REFERENCES:
- [Background] Amato PR, Booth A. The legacy of parents' marital discord: consequences for children's marital quality. J Pers Soc Psychol. 2001 Oct;81(4):627-38. PMID 11642350
- [Background] Arnett JJ. Emerging adulthood. A theory of development from the late teens through the twenties. Am Psychol. 2000 May;55(5):469-80. PMID 10842426
- [Background] Beach SR, O'Leary KD. Dysphoria and marital discord: are dysphoric individuals at risk for marital maladjustment? J Marital Fam Ther. 1993 Oct;19(4):355-68. doi: 10.1111/j.1752-0606.1993.tb00998.x. PMID 21118474